CLINICAL TRIAL: NCT02305147
Title: Etude Des Facteurs Prédictifs De L'apparition Et De L'évolution De La Maladie De Parkinson
Brief Title: Cohort Study to Identify Predictor Factors of Onset and Progression of Parkinson's Disease
Acronym: ICEBERG
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: IHU-A-ICM, Paris, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: C13-74
Record Dates: First submitted 2014-10-10; First posted 2014-12-02 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Biomarkers; Prognostic factors; Prodromal features; Disease progression
MeSH Terms: conditions — Parkinson Disease; Disease Progression | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sampling at baseline
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients with an idiopathic Parkinson Disease,: Patients with recent onset of Parkinson Disease: N=200
- Subjects at risk of PD: Subjects at risk to develop Parkinson Disease:
  * subjects with idiopathic Rem-sleep behavior disorder (iRBD): N=50
  * subjects related to a patient with genetically confirmed Parkinson Disease: N=30
  Interventions: Other: Clinical, biological and imaging followup
- Controls: Healthy controls: N=50
  Interventions: Other: Clinical, biological and imaging followup
- Patients with Parkinson Disease with genetic mutation: Patients with Parkinson Disease with a genetic mutation in parkin, LRRK2, SNCA or GBA (N=30)

INTERVENTIONS:
Other: Clinical, biological and imaging followup — Assessment of motor and non motor signs every 12 months. Imaging and blood, cerebral fluid, stools and skin samples for identification of biomarkers of disease phenotype and progression.
  Groups: Controls; Subjects at risk of PD

SUMMARY:
Observational, prospective, monocentric study to assess clinical features, imaging and biologic biomarkers in Parkinson disease (PD) patients and rate of progression compared to healthy controls (HC) and subjects at risk to develop PD.

The primary objective of this study is to identify clinical, imaging and biologic markers of PD onset and progression for use in clinical trials of disease-modifying therapies.

DETAILED DESCRIPTION:
ICEBERG will be a four-year natural history study of de novo idiopathic PD patients, healthy controls, and subjects at risk to develop PD (idiopathic Rem Behavior Disorder -iRBD, and probants of patients with PD genetically confirmed).

All subjects will be comprehensively assessed at baseline and every year thereafter. Subjects will undergo clinical (motor, neuropsychiatric, sleep, ocular and cognitive evaluations) and imaging assessments. Blood (including a DNA sample), stools, skin biopsy and cerebral spinal fluid (CSF) samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* All subjects: Male or female age 18 years and older, MMSE score > 26, negative pregnancy test in potentially child-bearing women (contraindication to SPECT with DatScan).
* Idiopathic Parkinson disease subjects: diagnosis confirmed according to UK Parkinson's Disease Society Brain Bank criteria (UKPDSBB); disease duration less than 3 years.
* Genetic Parkinson disease subjects: parkinson diagnosis confirmed and mutation in parkin, LRRK2, SNCA or GBA genes.
* Prodromal subjects: subjects with identified relative with PD genetically confirmed or subjects with diagnosis of idiopathic Rem sleep Behavior Disorder (iRBD); neurological examination normal (no signs of parkinsonism).
* Healthy subjects: neurological examination normal

Exclusion Criteria:

* All subjects: Psychiatric disorder or any progressive life-threatening disease, impairment precluding appropriate information and instructions given concerning participation to the study; contra-indication to MRI or SPECT scan.
* Parkinson disease subjects: no dopamine transporter deficit at SPECT scan; parkinsonism induced by neuroleptics; neuroleptics intake within 6 months; atypical parkinson syndrom (MSA, PSP, CBD...)
* Parkinson disease subjects with mutation in Parkin, LRRK2, SNCA or GBA gene: atypical parkinson disease syndromes due to either drugs (e.g., metoclopramide, flunarizine, neuroleptics) or metabolic disorders (e.g., Wilson's disease), encephalitis or degenerative diseases (e.g., progressive supranuclear palsy) or currently taking neuroleptics or has taken neuroleptics within 6 months of baseline or any biological anomaly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with recent onset of Parkinson Disease (less than 3 years since diagnosis) compared to subjects at risk to develop Parkinson Disease and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2014-11-06 (Actual); Primary Completion 2029-11-06 (Estimated); Study Completion 2029-11-06 (Estimated)

PRIMARY OUTCOMES:
Rates of change of clinical, imaging and biomic outcomes | 4 years (annual visits)
  Slopes of change of clinical, imaging and biomics compared between PD patients, subjects at risk to develop PD and healthy subjects.
  Identification of predictive factors of these rates of change. As examples, outcomes include: MDS-UPDRS, Mattis dementia rating scale, Non Motor Signs scale, DAT striatal uptake.

SECONDARY OUTCOMES:
Clinical milestones in PD patients | 4 years (annual visits)
  Occurence of complications such as falls, freezing, dyskinesias, motor fluctuations, cognitive impairment, dysautonomia.
  Identification of predictive factors of these complications. Rates of progression in sub-groups of patients defined by the presence of these complications.
Prodromal features in subjects at risk to develop PD | 4 years (annual visits)
  Prodromal features such as anosmia, dysautonomia, color vision impairment, will be evaluated at inclusion and during followup in subjects with iRBD or first-degree relatives of genetically confirmed PD patients.
  Frequency of these features will be compared between subjects who phenoconvert and those who don't.
  Relation between baseline DatSCAN binding and risk of phenoconversion will be analysed.
Phenoconversion in subjects at risk to develop PD | 4 years (annual visits)
  Phenoconversion is defined as occurence of an extrapyramidal syndrome, confirmed 12 months later.
  Exploratory analysis to determine whether rates of progression clinical, imaging and biomic markers may predict phenoconversion in groups of patients with iRBD or probants of patients with PD genetically confirmed.

CONTACTS AND LOCATIONS:
Overall Officials: Marie VIDAILHET, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, FRANCE; Jean-Christophe CORVOL, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris, FRANCE
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France